CLINICAL TRIAL: NCT00161759
Title: A Study to Assess the Safety and Efficacy of Fibrin Sealant (FS 4IU) for Wound Healing in Subjects With Burn Wounds Requiring Skin Grafting Procedures
Brief Title: Safety and Efficacy Study of Fibrin Sealant (FS 4IU) for Skin Graft Fixation and Wound Healing in Subjects With Burn Wounds
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 520001
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2006-10

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Fibrin Tissue Adhesive; Thrombin

INTERVENTIONS:
Drug: Sheet skin grafts affixed with Fibrin Sealant (lyophilized) with 4 IU/mL Thrombin

SUMMARY:
The purpose of this study is to assess if Fibrin Sealant 4IU is as safe and efficacious as staples (the current standard of care) to achieve fixation of skin grafts and wound healing in subjects with burn wounds. Each subject receives staples as well as FS 4IU on comparable treatment sites.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from either the subject or the subject's legally acceptable representative prior to screening activities
* Male or female age >= 6 and <= 65 years of age
* Total burn wounds measuring <= 40% TBSA to include a deep partial thickness/full thickness area requiring autologous split thickness sheet skin grafts
* The selected test area consisting of a contiguous, deep partial thickness/full thickness burn wound between 2% and 8% TBSA, which can be divided into two approximate halves or two bilateral wounds (each measuring between 1% and 4% TBSA)
* Females of child-bearing potential with a negative urine or serum pregnancy test on admission
* Able and willing to comply with the procedures required by the protocol

Exclusion Criteria:

* Conductive electrical burns and chemical burns
* Digits, head, genitalia, palms of hands, soles of feet, and face are excluded as test sites
* Circumferential burns are excluded as a test area
* 4th or 5th degree burns
* Test area with infection as determined clinically by the Investigator prior to surgery
* Venous or arterial vascular disorder directly affecting a designated test area
* Known immune deficiency disorder, either congenital or acquired
* Chronically malnourished as determined clinically by the investigator prior to surgery (Investigators are responsible for determining subjects are chronically malnourished during the screening process. Investigators should take into consideration the following parameters: Medical history and physical appearance, the subject's body mass index, and any significant laboratory findings)
* Severe respiratory problems or concurrent head trauma at hospital admission
* Any chronic condition requiring the use of systemic corticosteroids 30 days prior to study entry and anytime during the course of the study
* Known or newly diagnosed diabetics requiring insulin
* Any other acute or chronic concurrent medical condition(s) that in the Investigator's opinion are a contraindication to skin grafting and study participation
* Known or suspected hypersensitivity to bovine protein
* Concurrent participation in another clinical trial in which an investigational agent is used. (Subjects must not have been enrolled in another clinical trial within 30 days of enrolling in this trial).

Ages: 6 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2002-03; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Overall Officials: David G. Greenhalgh, MD, Principal Investigator — University of California Davis Medical Center, Sacramento; Shriners Hospitals for Children, Sacramento, CA; Marianne Cinat, MD, Principal Investigator — University of California Irvine, Orange, CA; Arnold Luterman, MD, Principal Investigator — University of South Alabama Medical Center, Mobile, AL; Nicole Gibran, MD, Principal Investigator — University of Washington Burn Center, Seattle, WA; Glenn D. Warden, MD, Principal Investigator — Shriners Hospitals for Children, Cincinnati, OH; David Herndon, MD, Principal Investigator — Shriners Hospitals for Children, Galveston, TX; Richard L. Gamelli, MD, Principal Investigator — Loyola University Medical Center, Maywood, IL; Sidney F. Miller, MD, Principal Investigator — Wright State University, Miami Valley Hospital, Dayton, OH; Daniel Lozano, MD, Principal Investigator — University of California, San Diego; Philip E. Fidler, MD, Principal Investigator — Bridgeport Hospital, Bridgeport, CT; Kevin Foster, MD, Principal Investigator — Maricopa Medical Center, Phoenix, AZ; William L. Hickerson, MD, Principal Investigator — Joseph M. Still Burn Center at Doctors Hospital, August, GA
Locations (12):
- United States (12):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Maricopa Medical Center, Phoenix, Arizona
  - UCI Medical Center, Orange, California
  - University of California Davis Medical Center; Shriners Hospitals for Children, Sacramento, California
  - UCSD Medical Center, San Diego, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Joseph M. Still Burn Center at Doctors Hospital, Augusta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Shriners Hospitals for Children, Cincinnati, Ohio
  - Wright State University, Miami Valley Hospital, Dayton, Ohio
  - Shriners Hospitals for Children, Galveston, Galveston, Texas
  - University of Washington Burn Center, Seattle, Washington